

### RESEARCH CONSENT FORM

Project Title: Randomized Control Trial of Buprenorphine vs Buprenorphine/naloxone on the

Effects of Maternal Symptomatology

**Department**: Department of Obstetrics, Gynecology, and Reproductive Medicine

You are being asked to be a volunteer in a research study.

### **PURPOSE**

Due to the widespread opioid epidemic, there are many pregnant women and new mothers who have experienced addiction and drug use over the course of their pregnancy. This study aims to compare buprenorphine (Subutex) versus buprenorphine/naloxone (Suboxone) in management of opioid use disorder in pregnancy. We expect to enroll approximately 132 pregnant women over a planned two year period to determine a difference between the two medications. However, to account for the possibility of up to a 10% drop out or loss to follow-up, the target enrollment of 72 for each of the groups (144 total pregnant women) is projected.

You are being asked to participate because you are a pregnant woman with a recent history of opioid use. We are attempting to determine if using either buprenorphine (Subutex) versus buprenorphine/naloxone (Suboxone) in pregnant women with opioid use disorders has a greater advantage in managing maternal withdrawal symptoms and drug cravings.

We will also gather information to compare outcomes of your pregnancy when taking buprenorphine (Subutex) versus buprenorphine/naloxone (Suboxone). This includes how weeks you are in pregnancy at delivery and if you deliver vaginally or by cesarean. Other information we will gather includes how well your baby does in the nursery and his or her length of stay in the hospital.

Your prenatal care and delivery of your baby will not be different whether or not you participate in this study. Medication-assisted treatment with either buprenorphine (Subutex) or buprenorphine/naloxone (Suboxone) requires a signed patient agreement before healthcare providers prescribe buprenorphine or buprenorphine/naloxone which is also not different whether you participate. Urine toxicology testing is also a routine part of care when caring for pregnant women receiving buprenorphine or buprenorphine/naloxone.

## **PROCEDURES**

## If you decide to be in this study, your part will involve:

- Completing a short questionnaire form about yourself
- Completing a drug craving questionnaire periodically throughout the pregnancy
- Assessments by your doctor periodically throughout the pregnancy
- Being randomly assigned (like the flip of a coin) to one of two groups:
  - Group 1: Taking daily buprenorphine throughout the pregnancy. You will receive the prescription for all the buprenorphine needed for your pregnancy and postpartum period.
  - Group 2: Taking daily buprenorphine/naloxone throughout the pregnancy. You will
    receive the prescription for all the buprenorphine/naloxone needed for your
    pregnancy and postpartum period.
- Provide urine samples for testing presence of drugs periodically during prenatal care.
- Giving a tablespoon of blood on the day you are admitted for delivery.
- Allowing a tablespoon of cord blood sampling at the time you deliver your baby.
- Allowing evaluation of your placenta, the afterbirth, following your delivery.
- Allowing study specimens to be used for future investigations.
- Allowing information to be gathered on your newborn including weight at delivery, Apgar scores, umbilical artery gas, admission to the neonatal intensive care unit (NICU) and number of days, neonatal complications such as difficulty breathing, infections, or overall complications, received morphine, neonatal abstinence syndrome

# **RISKS / DISCOMFORTS**

## The following risks/discomforts may occur as a result of you being in this study:

- You and your baby will be exposed to buprenorphine (Subutex) or buprenorphine/naloxone (Suboxone). Studies suggest that both buprenorphine and buprenorphine/naloxone use in pregnancy are safe; however, risks to the fetus and developing child are not completely known. We will be monitoring your urine for other drug use as we would do in all pregnancies we treat with buprenorphine.
- Your baby short-term effects from the medications may include developing withdrawal at birth and/or the first week of life. No clear long-term effects in the fetus have been identified from medication-assisted treatment with buprenorphine or buprenorphine/naloxone; however, risks to the developing child are not completely known. Based on other opioid medications, normal development is anticipated.
- Some women may occasionally experience withdrawal symptoms and drug cravings during this study as medications are being adjusted to ideal levels as per the usual protocol in women we treat with buprenorphine. Maternal withdrawal symptoms in pregnancy can also lead to withdrawal symptoms for your baby.
- Rarely some women may experience discomfort at the time of the blood draw. This may include temporary pain and bruising where the needle enters the skin, and sometimes, fainting and/or infection.
- There is a risk of allergic reaction to the buprenorphine or buprenorphine/naloxone

- Other common maternal adverse reactions include nausea, vomiting, diarrhea, headache, constipation, insomnia, rhinitis, diarrhea.
- Since this is a research study, not all risks may be known at this time; there may be unforeseen risks associated with study participation

### **BENEFITS**

- There may be no direct benefit to you if you decide to participate in the study.
- The study can provide indirect benefit to others through the information obtained about the use of buprenorphine or buprenorphine/naloxone in pregnancy.
- The information gained at the end of this study may help future healthcare providers in the management of opioid use disorder in pregnancy

**PAYMENT TO YOU** - You will not receive payment for taking part in the study.

### CONFIDENTIALITY

We will take steps to help make sure that all the information we get about you is kept confidential. Your name will not be used wherever possible. We will use a code instead. All the study data that we get from you will be kept locked up. The code will be locked up too. If any papers and talks are given about this research, your name will not be used.

We want to make sure that this study is being done correctly and that your rights and welfare are being protected. For this reason, we will share the data we get from you in this study with the study team and Stony Brook University's Committee on Research Involving Human Subjects, applicable Institutional officials, and certain federal offices, including the Office for Human Research Protections (OHRP), and, where applicable, the Food and Drug Administration (FDA). However, if you tell us you are going to hurt yourself, hurt someone else, or if we believe the safety of a child is at risk, we will have to report this.

In a lawsuit, a judge can make us give him the information we collected about you.

While you are in this study we will get data about you and your baby's health from the medical record. We will also get health data from the results of the tests you and the baby will have done in this study. You have a right to privacy but the data we get about your health in this study can be shared with the people referenced above (the study team, Stony Brook University's Committee on Research Involving Human Subjects, applicable institutional officials, and federal offices such as OHRP, FDA) as well as:

- your insurance company
- your medical doctor

You and your baby's health data are shared to make sure the study is being done correctly, costs are charged correctly, and to make sure your rights and safety are protected. Not all of these people are required by law to protect your health data. They might share it with others without your permission.

Some of the health information we get from you in this study, for example buprenorphine or buprenorphine/naloxone levels cannot be shared with you until the end of the study. Blood samples will be evaluated at the end of the study.

You have the right to stop allowing us to use or give out you or your baby's health data. You can do this at any time by writing to -----, MD. If you do this, we will stop collecting any new health data from you, except if we need to keep an eye on a bad side effect you were having in the study. We will use any data we collected before you wrote your letter. When you sign the consent form at the end, it means:

- That you have read this section.
- That you will allow the use and reporting of your health data as described above.
- You have received a form from the University Hospital. It is called the Notice of Privacy Practices form.

# **Clinical Trial Registry**

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## **COSTS TO YOU**

• There are no foreseeable costs to you.

### **ALTERNATIVES**

- Your alternative to being in this study is to simply not participate
- Seek medical treatment with an authorized methadone clinic or any other substance use disorder provider

## **IN CASE OF INJURY**

• If you are injured as a result of being in this study, please contact Dr. ---- at telephone (631) 444-7650. The services of Stony Brook University Hospital will be open to you in case of such injury. However, you and/or your insurance company will be responsible for payment of any resulting treatment and/or hospital stay.

## **CONSEQUENCES OF WITHDRAWING**

- If you decide to withdraw from the study, those in either group may discontinue medication use at any time.
- If you decide to withdraw from this study, the obstetric healthcare providers will continue to provide care to you through pregnancy and the postpartum period. Your medication-assisted treatment with buprenorphine or buprenorphine/naloxone will be continued

- unless the there is conflict with the patient agreement (similar if you not participating in this study)
- The consequence of stopping the medication without seeking alternate treatment can result in maternal withdrawal and drug craving side effects with potential to negatively affect the unborn baby.
- We recommend that if you decide to withdraw from this study, that you inform your primary obstetric healthcare provider or seek immediate medical attention with your primary doctor to receive adequate treatment to prevent unwanted side effects.

## **REMOVAL FROM STUDY**

• You may be removed from the study if you were chosen for the buprenorphine or buprenorphine/naloxone group but have not taken the prescribed medication as instructed, non-compliant to follow-up, medication is not effectively treating your symptoms, or if we decide to stop the study prematurely.

### YOUR RIGHTS AS A RESEARCH SUBJECT

- Your participation in this study is voluntary. You do not have to be in this study if you don't want to be.
- You have the right to change your mind and leave the study at any time without giving any reason, and without penalty.
- Any new information that may make you change your mind about being in this study will be given to you.
- You will get a copy of this a signed and dated copy of this consent form to keep.
- You do not lose any of your legal rights by signing this consent form.

### QUESTIONS ABOUT THE STUDY OR YOUR RIGHTS AS A RESEARCH SUBJECT

- If you have any questions, concerns, or complaints about the study, you may contact Dr. ----, at telephone # (631) 444-7650.
- If you have any questions about your rights as a research subject or if you would like to obtain information or offer input, you may contact -----, Committee on Research Involving Human Subjects, (631) 632-9036, OR by e-mail,----
- Visit Stony Brook University's Community Outreach page, <a href="http://www.stonybrook.edu/research/orc/community.shtml">http://www.stonybrook.edu/research/orc/community.shtml</a> for more information about participating in research, frequently asked questions, and an opportunity to provide feedback, comments, or ask questions related to your experience as a research subject.

If you sign below, it means that you have read (or have had read to you) the information given in this consent form, and you would like to be a volunteer in this study.

\_\_\_\_\_

| Subject Name (Printed) | Subject Signature | Date | Time |
|---|---|---|---|
| Name of Person Obtaining Consent (printed) | Signature of Person Obtaining Consent | Date | Time |